CLINICAL TRIAL: NCT02139462
Title: Optimizing Fidelity to Family-Based Treatment for Adolescent Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James Dale Lock, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R21MH096779-01 (NIH); SPO 103420 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Online Training for Therapists
Keywords: FBT, fidelity, training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard training (Experimental): Therapists will receive standard training in FBT.
  Interventions: Other: Standard FBT training
- Novel training (Experimental): Therapists will receive a novel, more efficient training in FBT
  Interventions: Other: Novel FBT training

INTERVENTIONS:
Other: Standard FBT training — Therapists will receive standard training in Family Based Treatment (FBT)
  Arms: Standard training
Other: Novel FBT training — Therapists will receive a novel training in Family Based Treatment (FBT)
  Arms: Novel training

SUMMARY:
This study will use a data base of archived therapy sessions of family therapy for adolescent anorexia nervosa to determine the role of fidelity to treatment and outcome. In addition, it will develop a novel, more efficient way to train therapists in family therapy for adolescent anorexia nervosa and examine if it is feasible to conduct a trial comparing this novel training to standard, more intensive training.

ELIGIBILITY:
Inclusion Criteria:

* masters or doctoral training in their field (psychology, psychiatry, family therapy).
* must be licensed
* have no reports of malpractice or loss of privileges at clinical institution
* minimum caseload 5 adolescents with AN each year over past 3 years
* no previous training in FBT
* computer/web access

Exclusion Criteria:

* Previous FBT training for AN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Feasibility | end of treatment (approximately 1.5 years after beginning training)
  The primary outcome will be feasibility (e.g., recruitment, attrition, assessment battery, resource costs) to conduct a sufficiently powered comparative study.

SECONDARY OUTCOMES:
Fidelity | Session 4, end of training (approximately 1.5 years after beginning training)
  Secondary outcomes include exploring differences in therapist fidelity and relationships between fidelity and patient outcomes between these two groups (e.g., fidelity and weight change at session 4).

CONTACTS AND LOCATIONS:
Overall Officials: James Lock, MD, PhD, Principal Investigator — Stanford University; Daniel Le Grange, PhD, Principal Investigator — University of California, San Francisco; W. Stewart Agras, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States